CLINICAL TRIAL: NCT04576377
Title: The Dynamics of the Immune Responses to Repeat Influenza Vaccination Exposures (DRIVE) Study - a Randomized Controlled Trial
Brief Title: Dynamics of the Immune Responses to Repeat Influenza Vaccination Exposures
Acronym: DRIVE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: University of Chicago (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BJC033; 1U01AI153700 (NIH)
Record Dates: First submitted 2020-09-29; First posted 2020-10-06 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — FluBlok

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Influenza vaccination (Experimental)
  Interventions: Biological: FluBlok
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: FluBlok — Recombinant HA quadrivalent influenza vaccine (0.5mL Flublok®, Sanofi Pasteur) containing 180μg antigen, 45μg for each influenza strain included.
  Arms: Influenza vaccination
Other: Placebo — 0.5mL saline placebo.
  Arms: Placebo

SUMMARY:
The aims of this vaccine trial are: (1) to measure humoral and selected cellular immune responses to repeated influenza vaccination with Flublok, including these responses' associations with age, birth year, and prior vaccination history; (2) to identify the characteristics of study participants who are vaccinated but still become infected with influenza virus ("vaccine failures") and participants who have poor immune responses to vaccination; and (3) to predict how influenza vaccinations and infections shape immunity.

DETAILED DESCRIPTION:
Background: Influenza vaccine is the most frequently used vaccine in the United States and globally. Influenza vaccination provides variable protection against influenza virus infection from year to year, with multiple factors contributing to variation in vaccine effectiveness. First, viral evolution necessitates regular updates to vaccine strains, and the degree of match between vaccine and circulating strains affects vaccine protection. A more serious issue, which motivates this study, is that repeated influenza vaccination may lead to "focusing" of immune responses to older strains, potentially reducing protection against recent strains.

Aims and objectives: The aims of this trial are: (1) to measure humoral and selected cellular immune responses to repeated influenza vaccination, including these responses' associations with age, birth year, and prior vaccination history; (2) to identify the characteristics of study participants who are vaccinated but still become infected with influenza virus ("vaccine failures"); and (3) to predict how influenza vaccinations and infections shape immunity.

Study design: *DRIVE I* A 4-year immunogenicity study with a randomized controlled design including 447 adults who are 18-45 years of age. Participants will be randomized to 5 groups in equal proportions, where the groups receive Flublok (Sanofi Pasteur) vaccine (V) or saline placebo (P) in years 1-4: group 1: V+V+V+V; group 2: P+V+V+V; group 3: P+P+V+V; group 4: P+P+P+V; group 5: P+P+P+P.

*DRIVE II* A 3-year and one-month immunogenicity study with a randomized controlled design among 530 adults who are 18-45 years of age. Participants will be randomized into 4 groups in equal proportions, where the groups will receive Flublok (Sanofi Pasteur) vaccine (V) or saline placebo (P) in year 1-4: group 1: V+V+V+V; group 2: P+V+V+V; group 3: P+P+V+V; group 4: P+P+P+V.

*DRIVE I & DRIVE II* All participants will receive influenza vaccination at the end of the final year. We will collect blood samples and nasal strip samples before vaccination and various timepoints after vaccination. Whole blood samples will be collected from a subset for later PBMC analysis. We will actively monitor participants for acute respiratory illnesses throughout the follow-up period, and collect and test respiratory swabs and blood samples to identify respiratory virus infections and acute immune responses to infection.

Number of Subjects: DRIVE I: 447 enrolled in autumn and winter 2020/21. DRIVE II: 530 enrolled in autumn and winter 2021/22.

Main outcome measures: The primary outcome measures are the humoral immune responses at day 30 after vaccination measured by hemagglutinin inhibition and microneutralization assays. The investigators will also study a number of secondary outcomes, including the persistence of immune responses 91, 182, 273 and 365 days after vaccination, and the immune responses to natural laboratory-confirmed influenza virus infections, as well as immunity and immune responses to other respiratory viruses including COVID-19 (SARS-CoV- 2).

Potential implications: Our study will provide novel insight into the effects of repeat influenza vaccination and infection on the strength and breadth of immune responses to influenza, the mechanisms underlying heterogeneity in vaccine response and vaccine failure, and biological factors that could explain variation in influenza vaccine effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years at enrolment.
* Capable of providing informed consent.
* Resident in Hong Kong in the coming 2 years.

Exclusion Criteria:

* Vaccinated against influenza in the past 24 months.
* Included in one of the priority groups to receive influenza vaccination in Hong Kong (priority groups include pregnant women, long-stay residents of institutions for persons with disability, persons with chronic medical problems (chronic cardiovascular, lung, metabolic or kidney diseases, obesity (body mass index 30 or above) and chronic neurological condition), healthcare workers or persons working in poultry, pig farming or pig slaughtering industry).
* With diagnosed medical conditions related to their immune system.
* Currently taking medication for any condition that impairs immune system.
* Individuals who report medical conditions not suitable to receive inactivated influenza vaccines, such as: Severe allergic reaction (e.g., anaphylaxis) after previous dose of any influenza vaccine; or to a vaccine component; moderate or severe acute illness with or without fever after any previous influenza vaccination; or a history of Guillain-Barré syndrome (GBS) within 6 weeks of previous influenza vaccination.
* Individuals, who report medical conditions not suitable to receive intramuscular injection, such as bleeding disorders; habitually taking anticoagulants (with the exception of antiplatelets such as aspirin).
* Individuals who have any medical conditions not suitable to receive inactivated influenza vaccines as determined by a clinician.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 977 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Immune response to vaccination (4-fold rise in titer at day 30) | 30 days after vaccination
  The proportion of participants who achieve a target rise in antibody titre against each of the vaccine strains at 30 days (the targeted rise in antibody titre is defined as the proportion of participants with a four-fold or greater rise in titer, i.e. either a pre-vaccination hemagglutination inhibition titer <10 and a post-vaccination hemagglutination inhibition titre ≥20, or a pre- vaccination hemagglutination inhibition titer ≥10 and at least a four-fold rise in post-vaccination hemagglutination inhibition antibody titer). The HAI assay has been unreliable for recent influenza A(H3N2) viruses, and if the vaccine strains or circulating strains in our study have this property we will use neutralization assays in place of HAI assays for the primary outcome for A(H3N2). Similarly, neutralization assays will be used if other influenza strains fail to hemagglutinate in the future.
Immune response to vaccination (GMT ratio at day 30 and 182) | 30 days and 182 days after vaccination
  The geometric mean titer (GMT) ratios between the vaccine group and the comparator group (placebo) against each of the vaccine strains at 30 days and 182 days

SECONDARY OUTCOMES:
Immune response to vaccination (antibody titer >=40 at day 30 and 182) | 30 days and 182 days after vaccination
  The proportion of participants who achieve an HAI titer ≥40 after each vaccination (or neutralization assay for H3N2 and any other non-hemagglutinating strains).
Immune response to vaccination (cell-mediated immunity) | 7 days and 30 days after vaccination
  The vaccine-induced influenza-specific CD4+ and CD8+ T cell responses 7 and 30 days post-vaccination, including cytokine production evaluated by Intracellular Cytokine Staining (ICS) assay. Responses for these and other relevant biomarkers are compared to the corresponding pre-vaccination values for each participant.
Immune response to vaccination (antibody specificity) | 30 days and 182 days after vaccination
  The fine-grained specificity and phenotypes of antibodies and influenza-positive B and T cell populations before and after vaccination and natural infection.
Incidence of reactions after vaccination [Safety] | 30 days after vaccination
  The rate of adverse events within 30 days after receipt of vaccination or placebo
Incidence of laboratory-confirmed influenza after vaccination (vaccine failure) | One year after vaccination
  The rate of polymerase chain reaction (PCR)-confirmed influenza virus infection.
Incidence of other respiratory infections | One year after vaccination
  The occurrence of other respiratory infections, including COVID-19 infections, in participants, determined by PCR or serology

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
We will release anonymized individual patient data along with publication of study results.
Supporting Information: Study Protocol, Analytic Code
Time Frame: On publication of study results
Access Criteria: Freely available on a public repository such as Dryad or Github

REFERENCES:
- [Derived] Cowling BJ, Wong SS, Santos JJS, Touyon L, Ort JT, Ye N, Kwok NKM, Ho F, Cheng SMS, Ip DKM, Peiris M, Webby RJ, Wilson PC, Valkenburg SA, Tsang JS, Leung NHL, Hensley SE, Cobey S. Preliminary Findings From the Dynamics of the Immune Responses to Repeat Influenza Vaccination Exposures (DRIVE I) Study: A Randomized Controlled Trial. Clin Infect Dis. 2024 Oct 15;79(4):901-909. doi: 10.1093/cid/ciae380. PMID 39041887